CLINICAL TRIAL: NCT03245736
Title: A Multi-center, Open-label Trial Investigating the Efficacy and Safety of Continued Treatment With Tisotumab Vedotin in Patients With Solid Tumors Known to Express Tissue Factor.
Brief Title: Tisotumab Vedotin Continued Treatment in Patients With Solid Tumors.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCT1015-03
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Ovary Cancer; Cervix Cancer; Endometrium Cancer; Bladder Cancer; Prostate Cancer; Esophagus Cancer; Lung Cancer, Nonsmall Cell; Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Esophageal Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — tisotumab vedotin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tisotumab Vedotin (Experimental): All patients will be administered tisotumab vedotin (HuMax-TF-ADC) in 21 day treatment cycles.
  Interventions: Drug: Tisotumab Vedotin

INTERVENTIONS:
Drug: Tisotumab Vedotin — All patients in the trial will be administered tisotumab vedotin (HuMax-TF-ADC).
  Other Names: TIVDAK

SUMMARY:
The purpose of the trial is to evaluate efficacy and safety of continued treatment with tisotumab vedotin.

DETAILED DESCRIPTION:
This is an open-label, multicenter trial to collect long-term safety and efficacy data and to provide ongoing access to tisotumab vedotin for patients with solid tumors who have completed a tisotumab vedotin base trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have either:

  1. completed the base trial and have shown a clinical benefit of SD or better and have never met any withdrawal criteria as defined in the tisotumab vedotin base protocol, or
  2. not completed treatment as defined in the base protocol for reasons that are not considered critical and unmanageable for the safety of the patient (as evaluated by the investigator and/or the sponsor) and the patient clearly showed response of PR or better.
* Patients must not have experienced radiographic disease progression or clinical signs of symptoms of instability requiring urgent intervention.
* Patients must not have received any other anti-cancer treatment (including surgery, radiation or systemic chemotherapy) since the base trial.
* Acceptable renal function
* Acceptable liver function
* Acceptable hematological status
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* A negative serum pregnancy test (if female and aged between 18-55 years old).
* Patients, both females and males, of reproductive potential must agree to use adequate contraception during and for six months after the last infusion of tisotumab vedotin.

  1. Adequate contraception for women is defined as hormonal birth control or an intrauterine device (safe hormonal contraceptives include contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release). In countries where two highly effective methods of contraception are required this will be an inclusion criterion.
  2. Male patients must be willing to use a latex condom during any sexual contact with females of childbearing potential during and for six months after the last infusion of tisotumab vedotin, even after having undergone a successful vasectomy.
  3. In order to be considered as sterilized or infertile, a patient must have undergone surgical sterilization (vasectomy/bilateral tubectomy; hysterectomy and bilateral ovariectomy) or be postmenopausal (12 months or more with no period prior to enrolment).
* Following receipt of verbal and written information about the trial, patients must provide signed informed consent before any trial-related activity is carried out.
* Acceptable coagulation status as defined in the applicable base protocol

  1. GEN701: Acceptable coagulation status: International normalized ratio (INR) ≤ 1.2 (without anticoagulant therapy), and activated partial thromboplastin time (aPTT) ≤ 1.25 ULN; patients on stable doses of therapeutic anti-coagulative treatment for ≥ 8 weeks (e.g., warfarin) must have an INR < 3.
  2. GEN702: Acceptable coagulation status defined as: INR ≤ 1.2 (without anticoagulant therapy), and aPTT ≤ ULN.

Exclusion Criteria:

* Presence of CTCAE (Common Terminology Criteria for Adverse Events) grade ≥ 2 peripheral neuropathy.
* Clinically significant active viral, bacterial or fungal infection requiring:

  1. Intravenous treatment with anti-infective therapy that has been administered less than two weeks prior to first dose in this trial, or
  2. Oral treatment with anti-infective therapy that has been administered less than one week prior to first dose in this trial.
  3. Prophylactic anti-infective therapy, which is given without clinical symptoms is allowed.
* Ongoing acute or chronic inflammatory skin disease.
* Women who are breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Genmab
Locations (4):
- Brian Slomovitz, Miami, Florida, United States
- United Kingdom (3):
  - Johann de Bono, Chelsea
  - Beatson Cancer Centre, Glasgow
  - Fiona Thistlethwaite, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants entered the trial following completion of other tisotumab vedotin trials such as GEN701 and GEN702. A total of 5 participants took part in the trial at 3 sites in the United Kingdom and 1 site in the United States from 23 August 2017 to 10 January 2019.
Pre-assignment Details: Six participants were screened, 5 of which were enrolled.
Groups:
- Tisotumab Vedotin: Tisotumab vedotin was administered as an intravenous (IV) infusion on Day 1 of each 21-day cycle (once every 3 weeks). The trial ran until the investigator determined that the participant was no longer benefiting from treatment (ie, disease progression or unacceptable toxicity had occurred), the trial was terminated by the sponsor, or the participant withdrew consent. Each participant received the same dose that they were exposed to in the previous base trial.
Period: Overall Study
Arm/Group | Tisotumab Vedotin
Started | 5
Completed | 0
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Progressive Disease | 4

BASELINE CHARACTERISTICS:
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 5
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 50.4 (10.46) [lower limit 10.46]
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0
  Preterm newborn infants (gestational age < 37 wks) | 0
  Newborns (0-27 days) | 0
  Infants and toddlers (28 days-23 months) | 0
  Children (2-11 years) | 0
  Adolescents (12-17 years) | 0
  Adults (18-64 years) | 5
  From 65-84 years | 0
  85 years and over | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Treatment Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical trial participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Treatment emergent adverse event (TEAE) is an AE occurring on or after the first dose of study medication or worsening during treatment period.
Time Frame: Day 1 to Week 24 plus 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 5
Participants | 5

2. Secondary Outcome: Objective Response Rate
Description: Objective Response was investigator-assessed based on the Response Evaluation Criteria In Solid Tumors version 1.1 [RECIST 1.1] criteria. The best overall response was reported for each participant.
Time Frame: Day 1 to Week 24 plus 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 5
Participants
  Complete Response | 0
  Partial Response | 2
  Stable Disease | 2
  Progressive Disease | 1

3. Secondary Outcome: Number of Participants With Increased Cancer Antigen (CA 125) Levels
Description: The number of participants with ovarian cancer whose levels of CA125 Antigen had increased since the end of the base trial are presented.
Time Frame: Day 1 to Week 24 plus 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 2
Participants | 1

4. Secondary Outcome: Number of Participants With Increased Prostate Specific Antigen (PSA)
Description: The number of participants with prostate cancer whose levels of PSA had increased since the end of the base trial are presented.
Time Frame: Day 1 to Week 24 plus 30 days
Population: No participants with prostate cancer participated in this trial.
Arm/Group | Tisotumab Vedotin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Week 24 plus 30 days
Groups:
- Overall: Tisotumab vedotin was administered as an intravenous (IV) infusion on Day 1 of each 21-day cycle (once every 3 weeks). The trial ran until the investigator determined that the participant was no longer benefiting from treatment (ie, disease progression or unacceptable toxicity had occurred), the trial was terminated by the sponsor, or the participant withdrew consent. Each participant received the same dose that they were exposed to in the previous base trial.
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=5)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=5)
Neuropathy peripheral (Nervous system disorders) | 4 (5)
Balance disorder (Nervous system disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Retinal exudates (Eye disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Localised infection (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 1 (3)
Ocular toxicity (Eye disorders) | 1 (1)
Corneal thinning (Eye disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Punctate keratitis (Eye disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed publications and presentations shall be submitted to the sponsor for its review at least 30 days before such presentation or publication is submitted to any third party.

DOCUMENTS (2):
  • Study Protocol (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/36/NCT03245736/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT03245736/SAP_001.pdf